CLINICAL TRIAL: NCT02361112
Title: A Phase I Study of Pyrotinib In Combination With Capecitabine In Patients With HER2 Positive Metastatic Breast Cancer
Brief Title: Study Evaluating Pyrotinib in Combination With Capecitabine In Patients With HER2 Positive Metastatic Breast Cancer
Acronym: BLTN-Ic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLTN-Ic
Record Dates: First submitted 2014-09-03; First posted 2015-02-11 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pyrotinib combined with capecitabine (Experimental)
  Interventions: Drug: pyrotinib combined with capecitabine

INTERVENTIONS:
Drug: pyrotinib combined with capecitabine

SUMMARY:
Pyrotinib is an oral tyrosine kinase inhibitor targeting both EGFR and HER-2 receptors. This study is designed to evaluate the safety and tolerability of Pyrotinib in combination with capecitabine in patients with HER2 positive metastatic breast cancer:

To evaluate the safety and tolerability of pyrotinib, and the maximum tolerated dose (MTD) To determine the dose-limiting toxicity (DLT) To determine the pharmacokinetic profile of Pyrotinib To assess preliminary antitumor activity To determine preliminary regimen dose for phase II study

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 and ≤70 years.
* ECOG performance status of 0 to 1.
* Life expectancy of more than 12 weeks.
* At least one measurable lesion exists.(RECIST 1.1)
* Histologically or cytologic confirmed HER2 positive metastatic breast cancer which failed prior therapies.
* No previous treatment of capecitabin during the past 1 year.
* Required laboratory values including following parameters:

ANC: ≥ 1.5 x 109/L Platelet count: ≥ 100 x 109/L Hemoglobin: ≥ 9.0 g/dL Total bilirubin: ≤ 1.5 x upper limit of normal, ULN ALT and AST: ≤ 1.5 x ULN BUN and creatine clearance rate: ≥ 50 mL/min LVEF: ≥ 50% QTcF: < 470 ms

* Signed informed consent.

Exclusion Criteria:

* Subjects with third space fluid that can not be controled by drainage or other methods.
* Steroid treatment for more than 50 days, or in need of long-term use of steroids.
* Subjects that are unable to swallow tablets, or dysfunction of gastrointestinal absorption.
* Less than 4 weeks from the last radiotherapy,chemotherapy，surgery，hermone treatment,target therapy, or less than 6 weeks from the nitrosoureas or mitomycin chemotherapy.
* Subjects with no efficacy during the previous treatment of capecitabine.
* Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry.
* Subjects who can not interrupt the using of the drugs that may cause QT prolongation during study.
* Subjects with intracranial lesions.
* Subjects with bone or skin as the only target lesion
* Treated or treating with HER2 tyrosine kinase inhibitors (TKIs) before study entry.
* Receiving any other antitumor therapy.
* Less than 4 weeks from the last clinical trial.
* Known history of hypersensitivity to pyrotinib、capecitabine or any of its components or metabolites.
* Ongoing infection (determined by investigator).
* History of immunodeficiency, including HIV-positive, suffering from other acquired, congenital immunodeficiency disease, or history of organ transplantation.
* Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial.
* Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test.
* Female patients of childbearing age that are reluctant to take effective contraceptive measures throughout the trial period.
* Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study. Examples include, but are not limited to,hypertension, severe diabetes, or thyroid disease.
* Alcoholism, smoking (daily ≥ 5 roots) and other bad habits.
* Known history of neurological or psychiatric disease, including epilepsy or dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one subject out of three experiences has a dose-limiting toxicity (DLT) upon completing one treatment cycle. | 21 days
  DLT was difined as the cetain AEs which were observed during the first cycle (D1-D21）of treatment.

SECONDARY OUTCOMES:
Cmax, Tmax, T1/2, AUCss and R of pyrotinib and capecitabine in combination | 12 months
the number of participants with adverse event | 12 months
preliminary antitumor activity for the regimen, objective response rate | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Guan X, Ma F, Li Q, Chen S, Lan B, Fan Y, Wang J, Luo Y, Cai R, Zhang P, Li Q, Xu B. Survival benefit and biomarker analysis of pyrotinib or pyrotinib plus capecitabine for patients with HER2-positive metastatic breast cancer: a pooled analysis of two phase I studies. Biomark Res. 2023 Feb 20;11(1):21. doi: 10.1186/s40364-023-00453-0. PMID 36803645
- [Derived] Li Q, Guan X, Chen S, Yi Z, Lan B, Xing P, Fan Y, Wang J, Luo Y, Yuan P, Cai R, Zhang P, Li Q, Zhong D, Zhang Y, Zou J, Zhu X, Ma F, Xu B. Safety, Efficacy, and Biomarker Analysis of Pyrotinib in Combination with Capecitabine in HER2-Positive Metastatic Breast Cancer Patients: A Phase I Clinical Trial. Clin Cancer Res. 2019 Sep 1;25(17):5212-5220. doi: 10.1158/1078-0432.CCR-18-4173. Epub 2019 May 28. PMID 31138588